CLINICAL TRIAL: NCT04711889
Title: Protective Effect of Ulinastatin Against Negative Inflammatory Response and Organ Dysfunction After Acute Type a Aortic Dissection Surgery (PANDA I)
Acronym: PANDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Hong Liu, Investigator of Nanjing Medical University, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PANDA I
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Acute Aortic Syndrome; Type a Aortic Dissection
Keywords: Acute Aortic Syndrome
MeSH Terms: conditions — Acute Aortic Syndrome | interventions — urinastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ulinastatin (Experimental): Ulinastatin 10 0000 Units is taken intravenously three times a day.
  Interventions: Drug: Ulinastatin
- Blank control (Sham Comparator): Blank control.
  Interventions: Drug: Blank control

INTERVENTIONS:
Drug: Ulinastatin — Ulinastatin is taken three times a day.
  Arms: Ulinastatin
Drug: Blank control — Blank control
  Arms: Blank control

SUMMARY:
Acute Aortic Syndrome (AAS) is a common feature of acute aortic wall events, including aortic dissection, intramural hematoma, aortic ulceration and aortic trauma, and occurs in up to 35 cases per 100,000 cases per year between the ages of 65 and 75 years. Ulinastatin has antiinflammatory activity and suppresses the infiltration of neutrophils and the release of elastase and chemical mediators from neutrophils. Recent studies have shown that ulinastatin may be cytoprotective against ischemia-reperfusion injury in the liver, kidney, heart, and lung. The authors aim to examine the association between decreased release of inflammatory response to urinary trypsin inhibitor treatment and decreased myocardial and lung injury after acute aortic syndrome surgery.

ELIGIBILITY:
Inclusion Criteria:

* The patients are conformed to 2010 ACC/AHA guidelines for the diagnosis and treatment of thoracic aortic disease (TAD) within two weeks of onset;
* Patients with type a acute aortic syndrome confirmed clinically and radiologically and planning to undergo aortic surgery were enrolled.
* The patients' age of 18 years or older.
* Agree to participate in the study and sign the informed consent.

Exclusion Criteria:

* Patients allergic to Ulinastatin;
* Lactating women and pregnant women;
* Patients with mental diseases;
* Refuse to participate in this study and refuse to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
SOFA score | mean SOFA score 7 days after surgery
  The daily SOFA score after baseline was calculated for each patient on the basis of organ systems: neurologic, cardiovascular, respiratory, renal, hepatic, and coagulation systems. (Scores for each system range from 0 to 4, with higher scores indicating more severe organ-system dysfunction)

SECONDARY OUTCOMES:
Mortality | 30 days after surgery
  Death from any cause

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The first affiliated hospital of nanjing medical university, Nanjing, Jiangsu
  - Beijing Anzhen Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Diao YF, Chen ZB, Gu JX, Xu XY, Lin WF, Yuan CZ, Xiong JQ, Li MH, Ni BQ, Zhao S, Shao YF, Zhang YY, Liu H. Incorporating Circulating Plasma Interleukin-10 Enhanced Risk Predictability of Mortality in Acute Type A Aortic Dissection Surgery. Rev Cardiovasc Med. 2025 Feb 21;26(2):26334. doi: 10.31083/RCM26334. eCollection 2025 Feb. PMID 40026520
- [Derived] Liu H, Qian SC, Zhu K, Diao YF, Xu XF, Tang ZW, Fan GL, Yue HH, Chen JQ, Yang JN, Zhang YY, Ma C, Liu X, Wu Y, Wu Z, Liu N, Li A, Ni BQ, Shao YF, Zhao S, Li HY, Zhang HJ; China Additive Anti-inflammatory Actions for Aortopathy and Arteriopathy (5A); PANDA Trial Investigators. Protective effect of ulinastatin against negative inflammatory response and organ dysfunction in acute aortic dissection surgery: The PANDA trial. Cell Rep Med. 2025 Jan 21;6(1):101888. doi: 10.1016/j.xcrm.2024.101888. PMID 39842406